CLINICAL TRIAL: NCT02256683
Title: Effects of Dabigatran in Patients With AF - A Prospective, Randomized, Open-label, Explorative, Blinded-endpoint Trial to Compare the Efficacy of Dabigatran With Phenprocoumon for the Resolution of LAA Thrombus in Patients With AF
Brief Title: Resolution of Left Atrial-Appendage Thrombus - Effects of Dabigatran in Patients With AF
Acronym: RE-LATED_AF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruiting problems
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Boehringer Ingelheim (Industry); Atrial Fibrillation Network (Other)
Responsible Party: Principal Investigator, Thomas Rostock, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-008; 2013-005364-26 (EudraCT Number)
Record Dates: First submitted 2014-09-12; First posted 2014-10-06 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation or Atrial Flutter; Thrombosis of Left Atrial Appendage
Keywords: atrial fibrillation; atrial flutter; Atrial-Appendage Thrombus; Thrombus resolution; Dabigatran; Phenprocoumon; Transesophageal Echocardiography
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Dabigatran; Phenprocoumon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dabigatran (Experimental): Dabigatran etexilate (Pradaxa®) 150 mg capsule by mouth twice daly for 3 up to 6 weeks depending on treatment response
  Interventions: Drug: Dabigatran etexilate
- Phenprocoumon (Active Comparator): Phenprocoumon (Marcumar®) 3 mg capsule by mouth according to INR (2-3) for 3 up to 6 weeks depending on treatment response
  Interventions: Drug: Phenprocoumon

INTERVENTIONS:
Drug: Dabigatran etexilate — After inclusion of the patients with LAA thrombus, they are treated according to the randomization either with Pradaxa® (150 mg bid) or Marcumar® (INR 2-3) for at least three weeks. Thrombus resolution will be determined by transesophageal echocardiography (TEE) 3 weeks after start of treatment and subsequently at week 4 and 6 if necessary, i.e. LAA thrombus has not yet resolved. The study is terminated for each patient with the resolution of the LAA thrombus or after 6 weeks of study treatment.
  Other Names: Pradaxa®
  Arms: Dabigatran
Drug: Phenprocoumon — After inclusion of the patients with LAA thrombus, they are treated according to the randomization either with Pradaxa® (150 mg bid) or Marcumar® (INR 2-3) for at least three weeks. Thrombus resolution will be determined by transesophageal echocardiography (TEE) 3 weeks after start of treatment and subsequently at week 4 and 6 if necessary, i.e. LAA thrombus has not yet resolved. The study is terminated for each patient with the resolution of the LAA thrombus or after 6 weeks of study treatment.
  Other Names: Marcumar®
  Arms: Phenprocoumon

SUMMARY:
The primary objective of this study is to assess whether Dabigatran leads to a faster complete left atrial appendage (LAA) thrombus resolution as compared to Phenprocoumon. The secondary objectives of this trial are to assess the impact of Dabigatran versus Phenprocoumon on complete LAA thrombus resolution rate until week 6 and change in LAA thrombus volume under treatment as well as to assess and compare safety and tolerability of both drugs. A total of 110 patients with atrial fibrillation and LAA thrombus will be randomized to receive either Dabigatran (150 mg bid) or Phenprocoumon (INR 2-3) for a least three weeks. Thrombus resolution will be determined by transoesophageal echocardiography (TEE) 3 weeks after start of study treatment and subsequently at week 4 and 6 if necessary, i.e. LAA thrombus has not yet resolved. The study is terminated for each patient with the resolution of the LAA thrombus. For those patients whose thrombus still exists after 6 weeks treatment, the study is also terminated. Further treatments will be decided at the discretion of the treating physician.

DETAILED DESCRIPTION:
BACKGROUND Dabigatran etexilate, a direct thrombin inhibitor and new oral anticoagulant (NOAC), has been shown to effectively prevent thromboembolic events in patients with atrial fibrillation (AF). However, there is a paucity of data on the antithrombotic efficacy and safety of dabigatran in the resolution of left atrial appendage (LAA) thrombi in AF patients.

OBJECTIVE The primary objective of the RE-LATED trial is to assess whether treatment with dabigatran results in a faster complete LAA thrombus resolution as compared to vitamin-K antagonist phenprocoumon. Secondary objectives are to assess the impact of dabigatran on complete LAA thrombus resolution rate during treatment of 6 weeks, and change in LAA thrombus volume under treatment. Furthermore, this study aims to assess and compare safety and tolerability of dabigatran vs. phenprocoumon.

METHODS The study is designed as a prospective, multicenter, randomized, open-label, controlled, explorative, blinded endpoint (PROBE) trial. Patients with AF and left atrial appendage thrombus confirmed by transesophageal echocardiography (TEE) will be randomized to receive either dabigatran (150 mg bid) or phenprocoumon (INR 2-3) for the resolution of LAA thrombus formation for at least 21 days. Thrombus resolution will be determined by TEE 3 weeks after treatment initiation and subsequently at week 4 and 6, if the primary study endpoint (LAA thrombus resolution) has not yet been achieved. A total of 110 patients are planned to get randomized.

CLINICAL CONTEXT This is the first controlled trial that investigates the safety and efficacy of a NOAC for the resolution of a LAA thrombus in patients with AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented non-valvular AF or atrial flutter (12-lead ECG)
* Newly diagnosed or confirmed LAA thrombus in TEE (time of detection ≤ 28 days)
* Patients 18 years old
* CHA2DS2-VASc Score 1
* CrCL 30 mL/min (Cockcroft-Gault)
* Women with childbearing potential have to practice a medically accepted contraception
* Ability of patient to understand the character and the individual consequences of the clinical trial
* Signed and dated informed consent before start of any specific trial procedures

Exclusion Criteria:

* Patients > 80 years
* Low body weight (< 50 kg)
* Previous failure of LAA thrombus resolution with a VKA or factor Xa antagonist
* Occurrence of LAA thrombus under long-term treatment (> 3 months) with vitamin K antagonists with an exception in the case of continued INR out of the target range
* Contraindications for oral anticoagulation therapy (see current Fachinformation for Pradaxa® (150 mg) and Marcumar® (3 mg))
* History of heart valve disorder (i.e., prosthetic valve or hemodynamically relevant valve disease)
* Valvular heart disease requiring intervention (including mechanical valves)
* Acute myocardial infarction or MI within the last 26 weeks
* Acute coronary syndrome (e.g. instable angina pectoris, STEMI, NSTEMI)
* Chronic Heart Failure (> NYHA IIIa)
* Previous haemorrhagic stroke
* TIA within the last 90 days
* Clinical relevant bleeding within the last 26 weeks
* Acute and subacute bacterial endocarditis
* Recurrent pulmonary embolism
* Esophagitis, gastritis and gastroesophageal reflux
* Thrombocytopenia or functional platelet defects
* Congenital or acquired coagulation or haemorrhagic disorders
* Liver diseases (liver enzymes >2 ULN)
* Renal insufficiency (CrCL below 30 mL/min)
* Pre-treatment with Dabigatran in doses higher than 110 mg bid
* Concomitant treatment with rivaroxaban, apixaban, and in case of approval during the course of the trial, also edoxaban
* Concomitant treatment with irreversible cyclooxygenase inhibitors (e.g. ASA) at doses > 100 mg/d.
* Concomitant treatment with high doses of Adenosine diphosphate (ADP) receptor inhibitors (e.g. clopidogrel) at doses > 75 mg/d
* Combined treatment with Adenosine diphosphate (ADP) receptor inhibitors (e.g. clopidogrel) and irreversible cyclooxygenase inhibitors (e.g. ASA) in any dose combination
* Planned treatment with long-term oral anticoagulants for alternative indications
* Concomitant treatment with P-glycoprotein (P-gp) inhibitors, i.e. verapamil.
* Need for continued treatment with ticlopidine, ticagrelor, prasugrel, systemic ketoconazole, itraconazole, posaconazole, cyclosporine, tacrolimus, dronedarone, rifampicin, phenytoin, carbamazepine, St. John's Wort or any cytotoxic/myelosuppressive therapy
* Concomitant treatment with medication not permitted
* Planned surgical intervention during expected study participation or previous surgical interventions within the last 30 days
* Other significant risk factors for bleeding complications (e.g. malignancy)
* Pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other clinical trials during the present clinical trial or within the last 90 days.
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Time to complete left atrial appendage (LAA) thrombus resolution | 3 up to 6 weeks
  Transoesophageal echocardiography (TEE) will be performed at screening and after three weeks of treatment. In case of persistence of the LAA thrombus after three weeks, study treatment will be continued for a maximum of further 3 weeks and the patients will undergo a TEE at weeks 4 and 6 for LAA thrombus assessment until LAA thrombus resolution can be confirmed. The study is finished for each patient with the resolution of the LAA thrombus. For patients with a thrombus persisting after 6 weeks treatment, the study will also be terminated.
  At each TEE examination existence of a LAA thrombus is documented (YES/NO).

SECONDARY OUTCOMES:
Complete LAA thrombus resolution until week 6 (yes/no) | 3 up to 6 weeks
  Transoesophageal echocardiography (TEE) will be performed at screening and after three weeks of treatment. In case of persistence of the LAA thrombus after three weeks, study treatment will be continued for a maximum of further 3 weeks and the patients will undergo a TEE at weeks 4 and 6 for LAA thrombus assessment until LAA thrombus resolution can be confirmed. The study is finished for each patient with the resolution of the LAA thrombus. For patients with a thrombus persisting after 6 weeks treatment, the study will also be terminated.
  At each TEE examination existence of a LAA thrombus is documented (YES/NO).
Change in LAA thrombus volume under treatment | 3 up to 6 weeks
  Transoesophageal echocardiography (TEE) will be performed at screening and after three weeks of treatment. In case of persistence of the LAA thrombus after three weeks, study treatment will be continued for a maximum of further 3 weeks and the patients will undergo a TEE at weeks 4 and 6 for LAA thrombus assessment until LAA thrombus resolution can be confirmed. The study is finished for each patient with the resolution of the LAA thrombus. For patients with a thrombus persisting after 6 weeks treatment, the study will also be terminated.
  If a LAA thrombus exists the longitudinal and transversal diameters (mm) in the 45-60° and in the 135° layer are measured.
  If a LAA thrombus exists based on the diameters the volume (mm3) of the LAA thrombus is calculated.
Occurrence of any adverse event | 3 up to 6 weeks
  Patient interview at each visit and at follow up phone call. In case of availability review of patients' health records.
Occurrence of major bleedings | 3 up to 6 weeks
  Patient interview at each visit and at follow up phone call. In case of availability review of patients' health records.
  Criteria for major bleedings in non-surgical patients:
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in haemoglobin level of 2.0 g/dl (1.24 mmol/l) or more, or leading to transfusion of two or more units of whole blood or red cells.
Occurrence of strokes (all-type, haemorrhagic, ischemic) ascertained by CCT or cMRT | 3 up to 6 weeks
  Patient interview at each visit and at follow up phone call. In case of availability review of patients' health records.
Occurrence of transient ischaemic attacks (TIAs) | 3 up to 6 weeks
  Patient interview at each visit and at follow up phone call. In case of availability review of patients' health records.
Occurrence of cardiovascular events requiring hospitalization | 3 up to 6 weeks
  Patient interview at each visit and at follow up phone call. In case of availability review of patients' health records.
Occurrence of other thromboembolic events | 3 up to 6 weeks
  Patient interview at each visit and at follow up phone call. In case of availability review of patients' health records.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rostock, MD, Principal Investigator — University Medical Center of the Johannes Gutenberg-University Mainz
Locations (14):
- Germany (14):
  - University Heart Center; Department of Cardiology and Angiology II, Bad Krozingen
  - Charité Universitätsmedizin Berlin, Berlin
  - Vivantes Clinical Center Am Urban; General Internal Medicine and conservative intensive care, Berlin
  - Klinikum Coburg GmbH, Coburg
  - University Heart Center; Department of Cardiology, Cologne
  - University Heart Center; Department of Invasive Electrophysiology, Dresden
  - University Heart Center; Department of Cardiology, Electrophysiology, Hamburg
  - Hannover Medical School; Department of Cardiology and Angiology, Hanover
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsmedizin Leipzig, Leipzig
  - University Hospital Mainz, II. Medical Clinic, Dept. of Electrophysiology, Mainz
  - University Medical Center, Münster
  - St. Vincenz-Hospital GmbH, Paderborn
  - Rostock University Hospital; Rhythmology and Clinical Electrophysiology, Rostock